CLINICAL TRIAL: NCT06381830
Title: Clinical Study of the Efficacy and Safety of Chimeric Antigen Receptor T-cell Therapy Following Autologous Stem Cell Transplantation for Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: Clinical Study of CAR-T Cell Therapy Following ASCT for R/R B-cell Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry); Suzhou Hongci Hematology Hospital, Suzhou, China (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASCT+CART
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Lymphoma, B-Cell; Autologous Stem Cell Transplantation
Keywords: Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma; CAR-T Cell Therapy; Autologous Stem Cell Transplantation
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Blood Component Removal; Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASCT+CAR-T (Experimental): Participants will receive autologous stem cell transplantation followed by chimeric antigen receptor T (CAR-T) cell therapy.
  Interventions: Other: Apheresis; Other: Autologous Stem Cell Transplantation; Drug: CAR-T Cell Therapy

INTERVENTIONS:
Other: Apheresis — Participants will undergo two separate apheresis procedures, including: G-CSF primed hematopoietic stem cell collection and peripheral blood mononuclear cell apheresis for CAR-T cell manufacturing.
Other: Autologous Stem Cell Transplantation — Participants are designed to receive myeloablative conditioning regimen prior to infusion of a minimum 2 x 10^6 CD34+ stem cells/kilogram.
Drug: CAR-T Cell Therapy — CAR-T cells will be infused within 7 days after autologous hematopoietic stem cell infusion (2-10×10^6 CAR-T/kg，ivgtt).
  Other Names: Chimeric Antigen Receptor T-cell

SUMMARY:
The study is designed to evaluate the efficacy and safety of chimeric antigen receptor T-cell therapy following autologous stem cell transplantation for relapsed/refractory B-cell Non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Chimeric antigen receptor T (CAR-T) cell therapy has emerged as a promising approach for relapsed or refractory B-cell Non-Hodgkin's lymphoma (R/R B-NHL), with a complete response (CR) rate of about 50%. It is also considered to be a reasonable consolidation option in low or unmeasurable disease states recently. Unfortunately, 40%-70% of patients experienced relapse after CAR-T cell therapy in the long-term follow up. Autologous stem cell transplantation (ASCT) with myeloablative chemotherapy can enhance the efficiency of CAR-T cells and alleviate tumor load, leading to a lower relapse rate. As a result, CAR-T cell therapy following ASCT may be a promising method for R/R LBCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years.
2. Pathological immunohistochemistry or flow cytometry confirmed that R/ R Large B-cell Non-Hodgkin's Lymphoma with measurable (the longest diameter greater than 1.5cm and the longest vertical diameter greater than 1.0cm) lesions.
3. Previously treated with 1 or more lines of therapy.
4. ECOG≤2#.
5. The main organ functions need to meet the following conditions:LVEF≥50%;CCr≥30 ml/min; ALT and AST≤3 times normal range.
6. Hematopoietic function needs to meet the following conditions: platelet count≥45×10^9/L; hemoglobin≥8.0 g/dL; absolute neutrophil count≥1.0×10^9/L.
7. Subjects of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study until the follow-up one year period of the study.
8. Estimated survival time ≥3 months.
9. Voluntary signing of informed consent and good compliance.

Exclusion Criteria:

1. Have used immunosuppressants or hormones within 2 weeks prior to apheresis, or have to use immunosuppressants or hormones after signing informed consent.
2. The presence of bacterial, fungal, viral, mycoplasma or other types of infection that, in the judgment of the investigator, are difficult to control.
3. Active hepatitis B or active hepatitis C.
4. HIV infection.
5. Have received CAR-T cell therapy or allogeneic hematopoietic stem cell transplantation prior to signing the informed consent.
6. Prior malignancy (other than Relapsed Refractory B-cell Non-Hodgkin's Lymphoma).
7. Pregnant or breasting-feeding women.
8. There is evidence of complications or medical conditions that could interfere with the conduct of the study or put patients at serious risk, including but not limited to serious cardiovascular disease.
9. Conditions deemed by the researchers to be inappropriate for participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 24 months
  Number of participants who will have achieved response after ASCT plus CAR-T cell Therapy.
Progression-free Survival（PFS） | Up to 24 months
  PFS is defined as the time from ASCT to progression, death or the last follow-up point

SECONDARY OUTCOMES:
Duration of Response(DOR) | Up to 24 months
  To measure the duration of response to ASCT Plus CAR-T Cell Therapy over a follow-up period of 24 months
Complete Response Rate | Up to 24 months
  Number of participants who will have achieved complete response after ASCT plus CAR-T cell Therapy.
Overall Survival（OS） | Up to 24 months
  OS will be assessed from ASCT plus CAR-T cell therapy to death or last follow-up.
Adverse events profile | Up to 24 months
  Number of participants with adverse events. Frequencies of toxicities based on the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Deipei Wu, M.D., Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China